CLINICAL TRIAL: NCT06184607
Title: Relationship of Distance Between Contact Point to Attachment Level With the Presence of Interdental Papilla in Maxillary Central Incisors: A Cross-sectional Study
Brief Title: Relationship Between Contact Point to Attachment Level and Presence of Interdental Papilla
Status: Recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Sakshi Perio
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Attachment Loss, Periodontal
MeSH Terms: conditions — Periodontal Attachment Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maxillary anterior interdental papilla: Presence or loss of interdental papilla with intact maxillary central incisors in systemically healthy patients
  Interventions: Other: Distance from contact point to attachment level

INTERVENTIONS:
Other: Distance from contact point to attachment level — A periodontal probe will be used to measure distance between contact point to attachment level in maxillary central incisors

SUMMARY:
Thorough search of literature revealed no study has correlated the presence/absence of papilla to the contact point to attachment level distance. It could be a non- invasive approach and there is no need to inject local anaesthesia to the patient. It might be beneficial in predicting the papilla reconstruction outcome in patient friendly and non-invasive way.

DETAILED DESCRIPTION:
The presence of interdental papilla specially of maxillary anterior tooth region is an essential esthetic component. Loss of papilla or black triangle is not appealing and it is concern for both patient and clinicians. Beside esthetic concern, black triangle is associated with phonetic problem and food impaction. Several factors which may influence the presence/absence of interdental papilla are alveolar bone height, gingival biotype, interdental space morphology, type of contact area. Different classification system to categorize interdental papilla loss have been proposed. In the landmark study by Tarnow, a correlation was found between vertical distance from contact point to bone crest and presence/ absence of interdental papilla. Interdental clinical attachment level may indirectly indicate the changes in underlying bone level and it has been proven to be an important prognostic factor in consideration of success of root coverage procedure. Thorough search of literature revealed no study has correlated the presence/absence of papilla to the contact point to attachment level distance. It could be a non- invasive approach and there is no need to inject local anaesthesia to the patient. It might be beneficial in predicting the papilla reconstruction outcome in patient friendly and non-invasive way.

ELIGIBILITY:
Inclusion Criteria:

* Intact maxillary central incisors
* Age 18-50 years
* Closed contact points
* No history of traumatic tooth injury
* Completion of cause related therapy before 3months
* Full mouth plaque score and full mouth bleeding score <15%

Exclusion Criteria:

* • Systemic ailments which affect periodontium

  * History of previous periodontal surgery
  * Tooth with a prosthetic crown or restoration involving cementoenamel junction (CEJ).
  * Pathologic tooth migration
  * Presence of cervical abrasion/erosions
  * Presence of dental caries in maxillary central incisors
  * Trauma from occlusion
  * Crowding or spacing in maxillary central incisors
  * Angular bone defects
  * Pregnant women
  * Mobile tooth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Systemically healthy patients with intact maxillary central incisors will be recruited from the outpatient department of Periodontics and Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
contact point-attachment level | 12 months
  A periodontal probe will be used to measure primary outcome measure
contact point-papilla tip | 12 months
  A periodontal probe will be used to measure primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sakshi Malhotra, MDS, Principal Investigator — PGIDS, Rohtak, Haryana
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No